CLINICAL TRIAL: NCT04400136
Title: Impact of Treatment With Protonic Pump Inhibitors After Laparoscopic Sleeve Gastrectomy on Gastro-esophageal Reflux Disease Symptoms: Pilot Study
Brief Title: PPI Therapy Impact on GERD After Sleeve Gastrectomy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Angelo Iossa, MD PhD, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: Lasapienza2020
Record Dates: First submitted 2020-05-13; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Gastro Esophageal Reflux; Barrett Esophagus; Bariatric Surgery Candidate
Keywords: reflux, PPI, sleeve gastrectomy
MeSH Terms: conditions — Gastroesophageal Reflux; Barrett Esophagus | interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP A - no PPI (No Intervention): no PPI treatment (control group)
- GROUP B PPI 1/day for 6 months (Experimental): (standard dose-long term): Lansoprazole oral tablets 30 mg once daily (before breakfast on an empty stomach) for 6 months
  Interventions: Drug: Lansoprazole oral tablets 30 mg
- GROUP C PPI 1/day for 3 months (Experimental): (standard dose-short term): Lansoprazole oral tablets 30 mg once daily (before breakfast on an empty stomach) for 3 months
  Interventions: Drug: Lansoprazole oral tablets 30 mg

INTERVENTIONS:
Drug: Lansoprazole oral tablets 30 mg — Post operative prescription
  Other Names: PPI tablet
  Arms: GROUP B PPI 1/day for 6 months; GROUP C PPI 1/day for 3 months

SUMMARY:
The trial would to try to establish:

* The best post-operative PPI prescription protocol after Sleeve Gastrectomy
* The impact of PPI therapy on postoperative peptic diseases (erosive gastropathies, ulcers, duodenitis, esophagitis and/or Barrett)
* The impact of PPI therapy on post-operative GERD symptoms (assessed with the use of two standard tests: MRGE-HRQL and GERDQ

DETAILED DESCRIPTION:
45 patients candidate to primary SG and randomized in 3 study groups (15 per group) GROUP A: no treatment (control group)

GROUP B (standard dose-long term): Lansoprazole buccal tablets 30 mg once daily (before breakfast on an empty stomach) for 6 months

GROUP C (standard dose-short term): Lansoprazole buccal tablets 30 mg once daily (before breakfast on an empty stomach) for 3 months

ELIGIBILITY:
Inclusion Criteria:

* Patients candidates for primary SG
* Patients adhering to the follow-up protocol
* Age between 18 and 65 years
* No BMI limits

Exclusion Criteria:

* Gastric and/or esophageal diseases (routine preoperative endoscopy)
* Patients candidate for revisional bariatric surgery
* Chronic preoperative PPI therapy
* Using of PPI treatment for postoperative complications
* Conversion to open surgery
* Patients allergic to PPI
* Patients undergoing concomitant surgery
* Patients with hiatal hernia undergoing concomitant cruroplasty

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of post-operative GERD based on the trial protocol. Clinical evaluation | 12 months
  Questionnaire evaluation (GERD-HRQL score from 0 (no symptoms) to 5 (symptoms worsening daily activity) and GERD-Q (score A <8 no GERD, score A >8 and B > 3 GERD worsening normal life)

SECONDARY OUTCOMES:
evaluate in each group of the study (arm type) the endoscopic finding of peptic lesions of the esophagus-gastro-duodenal mucosa at 24 months of follow-up | 24 months
  Mucosal damage evaluation and stratified accordingly

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rome "la sapienza", Latina, Italy